CLINICAL TRIAL: NCT03852225
Title: Correlation Between End-tidal CO2 and Degree of Compression of Heart Cavities Measured by Transthoracic Ultrasound During Cardiopulmonary Resuscitation for Out-of-hospital Cardiac Arrest
Brief Title: Correlation Between End-tidal CO2 and Degree of Compression of Heart During CPR Measured by Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Roman Skulec, MD, PhD, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Other Study IDs: 2018-02
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cardiopulmonary Resuscitation; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA patients: Patients resuscitated for out-of-hospital cardiac arrest of non-traumatic origin and investigated by intra-arrest echocardiography.
  Interventions: Diagnostic Test: Intra-arrest echocardiography

INTERVENTIONS:
Diagnostic Test: Intra-arrest echocardiography — Intra-arrest echocardiography performed by portable ultrasound device during ongoing chest compressions.

SUMMARY:
Individual optimization of cardiopulmonary resuscitation (CPR) in real time may increase the success rate of the procedure. End-tidal CO2 (EtCO2) levels reflect cardiac output induced by CPR. Other potential marker of haemodynamic efficacy of CPR is direct measurement of the extent of induced compression of left ventricle (LV), right ventricle (RV) and inferior caval vein (IVC) by ultrasound. We plane to evaluate whether these ultrasound parameters correlate with EtCO2 levels during CPR for out-of-hospital cardiac arrest (OHCA) of non-traumatic origin.

DETAILED DESCRIPTION:
Pre-hospital observational study will be realized in the setting of physician-based Emergency Medical System in the Czech republic. 20 patients resuscitated for OHCA of nontraumatic origin are planned to be included to the study. Transthoracic echocardiography will be performed from subcostal view during ongoing chest compressions in all of them and in the time of this investigation EtCO2 level will be recorded. This will be repeated three times during CPR in each patient if possible. Later on, maximal and minimal diameter of LV, RV and IVC will be obtained from the recorded loops and compression index (%) of LV (LVCI), RV (RVCI) and IVC (IVCCI) will be calculated as (maximal-minimal/maximal cavital diameter)x100. Correlations between EtCO2 and LVCI, RVCI and IVCI and CImax will be expressed as Spearman's correlation coefficient.

The results of the study will answer the question whether echocardiographic evaluation of compression of heart cavities during CPR reflect haemodynamic efficacy of CPR. If so, this study will be followed by an interventional clinical trial evaluating the effect of compression depth changes as a response to measured compression of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient resuscitated for out-of-hospital cardiac arrest of non-traumatic origin.

Exclusion Criteria:

* Technical unavailability of intra-arrest ultrasonography and capnography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients meeting inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of EtCO2 level and compression index of left ventricle, right ventricle and inferior caval vein | Participant will be repeatedly evaluated during cardiopulmonary resuscitation. Therefore, anticipated time frame the time interval will fluctuate from 5 minutes to 120 minutes
  Compression index of left ventricle, right ventricle and inferior caval vein measured by intra-arrest echocardiography and EtCO2 measured by side stream approach during cardiopulmonary resuscitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency Medical Service of the Central Bohemian Region, Kladno, Central Bohemia, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skulec R, Vojtisek P, Cerny V. Correlation between end-tidal carbon dioxide and the degree of compression of heart cavities measured by transthoracic echocardiography during cardiopulmonary resuscitation for out-of-hospital cardiac arrest. Crit Care. 2019 Oct 29;23(1):334. doi: 10.1186/s13054-019-2607-2. PMID 31665061